CLINICAL TRIAL: NCT01778023
Title: A 12-month, Open-labelled, Randomised, Parallel-group, Multi-centre, Interventional Trial to Evaluate the Efficacy and Safety of Recombinant Human Growth Hormone (hGH) (Norditropin® Nordilet®) Therapy on Height Velocity (Ht-V) in Patients With Idiopathic Short Stature in Korea
Brief Title: Efficacy and Safety of Recombinant Human Growth Hormone on Height Velocity in Subjects With Idiopathic Short Stature
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GH-3899; U1111-1125-4790 (Other: WHO); 2015-002613-30 (EudraCT Number)
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Growth Disorder; Idiopathic Short Stature
MeSH Terms: conditions — Growth Disorders | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hGH:12months treatment (Experimental)
  Interventions: Drug: somatropin
- hGH: 6 month un-treatment + 6 month treatment (Active Comparator)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — A weekly dosage of 0.469 mg of somatropin per kg of body weight per week will be injected subcutaneously (under the skin) in the evening in 7 days per week.

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to evaluate the efficacy and safety of recombinant human growth hormone (hGH) in subjects with idiopathic short stature in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from subject's parents or legally acceptable representative before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject.)
* Pre-pubertal status (males aged from 4 to 11 [both inclusive], females aged from 4 to 9 [both inclusive]): an absence of breast development in females (Tanner 1 only) and testicular volume below 4 mL in males
* Growth hormone level above 10 ng/mL following a stimulation test (test result within 6 months from screening can be used)
* Height below 3 percentile
* Bone age below or equal to 12 year
* Epiphyses confirmed as open in patients at least 10 years or more of age

Exclusion Criteria:

* Known presence of one or more pituitary hormone deficiencies (ACTH (adrenocorticotropic hormone), ADH (antidiuretic hormone), FSH (follicle-stimulating hormone), LH (luteinising hormone), TSH (thyroid-stimulating hormone))
* Known primary hypothyroidism, adrenal insufficiency or hypogonadism (treated or untreated)
* Specific types of growth failure including, but not limited to, known chromosomal abnormalities associated with growth failure and altered sensitivity to growth hormone
* Bone age is advanced over chronological age more than 3 years
* Active malignancy, CNS (central nervous system) trauma, active chemotherapy or radiation therapy for neoplasia
* Prior history of intracranial hypertension
* Hypertrophic cardiomyopathy

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2013-01-17 (Actual); Primary Completion 2014-12-17 (Actual); Study Completion 2014-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (4):
- South Korea (4):
  - Novo Nordisk Investigational Site, Busan
  - Novo Nordisk Investigational Site, Daegu
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Suwon

REFERENCES:
- [Result] Safety and Efficacy Evaluation of Human Growth Hormone (GH) Therapy in Patients with Idiopathic Short Stature (ISS) in Korea - a Randomized Controlled Trial; Min Ho Jung, Byung-Kyu Suh, Cheol Woo Ko et al.; 028-042-GH-Pediatrics (posters) ENDO meeting 2016, Boston Massachusetts
- [Derived] Jung MH, Suh BK, Ko CW, Lee KH, Jin DK, Yoo HW, Hwang JS, Chung WY, Han HS, Prusty V, Kim HS. Efficacy and Safety Evaluation of Human Growth Hormone Therapy in Patients with Idiopathic Short Stature in Korea - A Randomised Controlled Trial. Eur Endocrinol. 2020 Apr;16(1):54-59. doi: 10.17925/EE.2020.16.1.54. Epub 2019 Oct 15. PMID 32595770
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 10 sites in Korea.
Groups:
- Group A: 12-month GH Treatment: For 12 months, a weekly dosage of 0.469 mg of somatropin (hGH) per kg of body weight was injected subcutaneously in the evening in seven (7) days per week using the Norditropin® Nordilet®.
- Group B: 6-month Untreated + 6-month GH Treatment: Subjects participated in the trial for 12 months. For the first six months of the trial period, subjects were untreated. For the last six months of the trial period, a weekly dosage of 0.469 mg of somatropin (hGH) per kg of body weight was injected subcutaneously in the evening in seven (7) days per week using the Norditropin® Nordilet®.
Period: Overall Study
Arm/Group | Group A: 12-month GH Treatment | Group B: 6-month Untreated + 6-month GH Treatment
Started | 36 | 18
Exposed | 36 | 15
Completed | 36 | 15
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: 12-month GH Treatment | Group B: 6-month Untreated + 6-month GH Treatment | Total
Number analyzed (Participants) | 36 | 15 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.3 (1.5) | 5.9 (1.2) | 6.2 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 6 | 23
  Male | 19 | 9 | 28
Height [Mean (Standard Deviation); unit: cm] — N=32, 15 due to missing baseline values for this characteristics.
  cm | 107.7 (8.7) | 105.8 (7.5) | 107.1 (8.3)

OUTCOME MEASURES:

1. Primary Outcome: Height Velocity (Ht-V)
Description: Height velocity (Ht-V) (cm/year) is the change in height per year (after 6 months of treatment). Ht-V was calculated by Novo Nordisk.
Time Frame: After 6 months of treatment
Population: Full analysis set (FAS) - included all randomised subjects in Group A who received at least one dose of the trial product and all randomised subjects in Group B. Four (4) subjects had missing height at baseline visit.
Measure: Least Squares Mean (Standard Error); unit: cm/year
Arm/Group | Group A: 12-month GH Treatment | Group B: 6-month Untreated + 6-month GH Treatment
Number analyzed (Participants) | 32 | 15
cm/year | 12.02 (0.29) | 6.87 (0.43)
Statistical Analysis 1: Comparison: Group A: 12-month GH Treatment vs Group B: 6-month Untreated + 6-month GH Treatment; Let D be a mean difference of the primary endpoint between group A and group B. Null hypothesis H0: D = 0 vs. alternative H1: D ≠ 0 will be statistically tested by an ANOVA model; Test type: Superiority or Other; p < 0.0001, ANOVA; The HV after 6 months of treatment was analysed using an ANCOVA method with group and sex as fixed effects, and age as a covariate; Treatment Difference = 5.15, 95% CI 2-sided [4.09 to 6.21]

2. Secondary Outcome: Change in Ht-SDS (Height Standard Deviation Score)
Description: Height standard deviation scores (HSDS) were calculated using Korean growth data (reported by the Korea Centre for Disease Control and Prevention). The mean normal range for HSDS is from -2 to +2. Negative scores below -2 indicate a height below normal range, whereas positive scores above +2 indicate a height above normal.
Time Frame: After 6 months of treatment.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Standard Deviation Score (SDS)
Arm/Group | Group A: 12-month GH Treatment | Group B: 6-month Untreated + 6-month GH Treatment
Number analyzed (Participants) | 32 | 15
Standard Deviation Score (SDS) | 0.76 (0.04) | 0.19 (0.06)

3. Secondary Outcome: Change in IGF Related Factors: IGF-I (Insulin-like Growth Factor-I)
Description: IGF-I (insulin-like growth factor-1) was measured at Visit 1 (screening),Visit 3 (3 months ± 7 days ),Visit 4 (6 months ± 7 days),Visit 5 (9 months ± 7 days ) and Visit 6 (12 months ± 7 days ). Change of IGF-I from baseline to 6 months treatment was calculated.
Time Frame: After 6 months of treatment.
Population: Full analysis set (FAS) - included all randomised subjects in Group A who received at least one dose of the trial product and all randomised subjects in Group B.
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | Group A: 12-month GH Treatment | Group B: 6-month Untreated + 6-month GH Treatment
Number analyzed (Participants) | 36 | 15
ng/ml | 192.58 (14.00) | 28.03 (21.81)

4. Secondary Outcome: Change in IGF Related Factors: IGFBP-3 (Insulin-like Growth Factor Binding Protein-3)
Description: IGFBP-3 was measured at Visit 1(screening), Visit 3 (3 months ± 7 days ), Visit 4 (6 months ± 7 days), 5 (9 months ± 7 days ) and 6 ( 12 months ± 7 days). Change of IGFBP-3 from baseline to 6 months treatment were calculated.
Time Frame: After 6 months of treatment.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mcg/mL
Arm/Group | Group A: 12-month GH Treatment | Group B: 6-month Untreated + 6-month GH Treatment
Number analyzed (Participants) | 36 | 15
mcg/mL | 0.89 (0.19) | 0.22 (0.30)

5. Secondary Outcome: Change in Bone Age
Description: Change in bone age from the baseline to 6 months.
Time Frame: After 6 months of treatment.
Population: Safety analysis set (SAS) :includes all subjects in Group A receiving at least one dose of the trial product and all subjects in Group B who had any available data after Visit 2.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Group A: 12-month GH Treatment | Group B: 6-month Untreated + 6-month GH Treatment
Number analyzed (Participants) | 36 | 15
years | 0.5 (0.2) | 0.5 (0.2)

6. Secondary Outcome: Occurrence of Adverse Events
Description: AEs were collected throughout the trial in both groups.
Time Frame: Throughout the trial (12 months)
Population: Safety analysis set - includes all subjects in Group A receiving at least one dose of the trial product and all subjects in Group B who had any available data after Visit 2.
Measure: Number; unit: events
Arm/Group | Group A: 12-month GH Treatment | Group B: 6-month Untreated + 6-month GH Treatment
Number analyzed (Participants) | 36 | 15
events | 70 | 25

7. Secondary Outcome: Ht-V (Height Velocity)
Description: Height velocity (Ht-V) (cm/year) is the change in height per year (after 6 months of treatment). Three sort of Ht-V was calculated from height data at Visit 2 (day 0), 4 (6 months ± 7 days) and 6 (12 months ± 7 days), as follows: Between Visits 2 and 4, between Visit 4 and 6 and between Visit 2 and 6. Ht-V was calculated by Novo Nordisk. It is the difference between Ht-V for the last 6 months and Ht-V for the first 6 months of treatment. This endpoint was only evaluated for Group A as per the trial protocol.
Time Frame: At the first 6 months and the last 6 months in group A
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: cm/year
Arm/Group | Group A: 12-month GH Treatment
Number analyzed (Participants) | 32
cm/year | 2.80 [1.55 to 4.04]

ADVERSE EVENTS:
Description: Safety analysis set - includes all subjects in Group A receiving at least one dose of the trial product and all subjects in Group B who had any available data after Visit 2.
Arm/Group | Group A: 12-month GH Treatment | Group B: 6-month Untreated + 6-month GH Treatment
Serious Adverse Events (participants affected / at risk) | 4/36 | 2/15
Other Adverse Events (participants affected / at risk) | 20/36 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: 12-month GH Treatment (N=36) | Group B: 6-month Untreated + 6-month GH Treatment (N=15)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Kawasaki's disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: 12-month GH Treatment (N=36) | Group B: 6-month Untreated + 6-month GH Treatment (N=15)
Eye disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 15 (43) | 7 (14)
Rhinitis (Infections and infestations) | 0 (0) | 2 (3)
Upper respiratory tract (Infections and infestations) | 3 (3) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to not release data until specified milestones, e.g. when the clinical trial report is available. At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.